CLINICAL TRIAL: NCT02454764
Title: To Study the Efficacy of 'Tenofovir Pulse and Peg Interferon Alpha 2b' Therapy in HBeAg-positive Patients With Normal ALT - A Randomized Control Trial
Brief Title: 'Tenofovir Pulse and Peg Interferon Alpha 2b' Therapy in HBeAg-positive Patients With Normal ALT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HBV-001
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2016-07

CONDITIONS: HBV
MeSH Terms: interventions — Tenofovir; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir + Interferon alpha 2 b (Experimental)
  Interventions: Drug: Tenofovir disoproxil Fumarate
- Tenofovir (Active Comparator)
  Interventions: Drug: Tenofovir + Interferon alpha 2b

INTERVENTIONS:
Drug: Tenofovir + Interferon alpha 2b
  Arms: Tenofovir
Drug: Tenofovir disoproxil Fumarate
  Arms: Tenofovir + Interferon alpha 2 b

SUMMARY:
After fulfillment of the selection criteria, all the patients included in the trial will be administered Tenofovir that will be continued for 3 months and then stopped for 1 month, LFT's, HBV DNA, HBsAg, will be checked weekly during the time period of stopping Tenofovir and thereafter at 4 months patients with ALT >/= 1.5 times ULN will be randomised in 2 groups to administer either Peg INF alpha 2b + Tenofovir (in same dose as before) or Tenofovir alone which will be continued for 48 weeks and the patients with no rise in ALT will be excluded. Patients will be closely monitored during the period of stopping tenofovir post pulse therapy and liver function tests will be performed weekly. Patients will be closely observed for the development of acute hepatitis or decompensation during the 4 - week period of drug withdrawal. Thereafter, CBC, KFT, LFT's, PT-INR, HBsAg (Q), HBeAg and HBV DNA levels will be tested every 3 months. After stopping treatment followup will be done at 24 weeks post stoppage of treatment to look for sustained seroconversion and virological/biochemical response

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naive chronic HBV infection i.e detectable HBsAg for past 6 months,
2. HBeAg (+),
3. ALT < ULN (Upper Limit Normal) on 2 or more occasions in last 6 months [ULN: 45]
4. HBV DNA >2000 IU/mL
5. Age > 18 years

Exclusion Criteria:

1. Decompensated Cirrhosis
2. Severe HBV flare with reactivation
3. Presentation as ACLF (Acute on Chronic liver Failure)
4. Baseline ALT > ULN (Upper Limit Normal)
5. Contraindications to PEG-IFN therapy
6. Prior HBV antiviral therapy within 6 months of enrollment
7. Co-infections with HCV/HIV
8. ANA +(autoantibodies suggestive of autoimmune disease) >1:80
9. Patient not willing for enrollment in the study
10. Pregnancy, lactation
11. Patients who leave the study/ discontinue the therapy before completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Sustained [ 6 months after stopping treatment] HBeAg seroconversion to anti-Hbe on two consecutive assays, at least 1 month apart | 65 weeks

SECONDARY OUTCOMES:
HBsAg loss | 64 weeks
Absence of quantifiable serum HBV DNA | 64 weeks
Development of serious adverse effects, acute hepatitis or hepatic decompensation | 64 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India